CLINICAL TRIAL: NCT05535569
Title: Phase Ib/II Study to Evaluate the Safety and Efficacy of Nivolumab in Combination With Paclitaxel in Epstein-Barr Virus(EBV)-Related, or Microsatellite Instability-High (MSI-H), or Programmed Cell Death Ligand 1 (PD-L1) Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0277
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Recurrent/Metastatic Gastric Cancer
Keywords: Epstein-Barr Virus(EBV)-Related, or Microsatellite Instability-High (MSI-H), or Programmed Cell Death Ligand 1 (PD-L1) Positive Advanced Gastric Cancer; Nivolumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Nivolumab, Paclitaxel

INTERVENTIONS:
Drug: Nivolumab, Paclitaxel — Increasing dose levels of paclitaxel (70 mg/m2 or 80 mg/m2 on Days 1, 8 and 15 of a 28-day treatment cycle) in combination with a fixed dose of nivolumab (3 mg/kg on Days 1 and 15 of a 28-day treatment cycle) will be explored using a 3+3 design to evaluate the safety and tolerability and to determine a MTD.

SUMMARY:
This is a Phase Ib/II study to identify the recommended dose of paclitaxel and nivolumab for further study, and to assess the safety and clinical efficacy of this combined treatment in EBV-related, MSI-high, or PD-L1 positive advanced gastric cancer after first line treatment.

DETAILED DESCRIPTION:
This is a Phase Ib/II study to identify the recommended dose of paclitaxel and nivolumab for further study, and to assess the safety and clinical efficacy of this combined treatment in EBV-related, MSI-high, or PD-L1 positive advanced gastric cancer after first line treatment.

Patients who are EBV-related, MSI-high, or PD-L1 positive will be confirmed by immunohistochemistry (IHC) in a central laboratory (Yonsei Cancer Center), and who meet all eligibility criteria will be enrolled to this study and receive treatment with nivolumab and paclitaxel until progressive disease is confirmed or at least 1 discontinuation criterion is met. It was assumed that about 15% of screened patients will be categorized EBV-related, MSI-high, or PD-L1 positive gastric cancer based on previously reported study results. Part 1>> Phase Ib Phase Ib: 6-12 (The actual number of subjects will be determined by the number of dose escalations to identify MTD and RP2D) Part 2>> Phase II - At the RP2D dose level in phase I part, we will expand phase 2 study for a total of 50 patients. Patients will be treated until the time of disease progression, intolerable toxicities, patient's refusal or consent withdrawal. Tumor assessment will be done every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided digned written informed Consent
2. Is male or female ≥19 years of age
3. Has a histologically or cytologically confirmed diagnosis of advanced gastric adenocarcinoma
4. Has documented EBV-related, MSI-high, or PD-L1 positive tumor in primary or metastatic tumor tissue
5. Has a life expectancy of at least 3 months
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Has measurable or evaluable disease as determined by RECIST 1.1.
8. Is able to swallow and retain orally administered medication
9. Has an adequate baseline organ function defined as:

   * White blood cells ≥3000/mm3 and neutrophils ≥1500/mm3
   * Platelets ≥100000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 × upper limit of normal (ULN) of the study site (or ≤5.0 × ULN in patients with liver metastases)
   * Total bilirubin ≤2.0 × ULN
   * Creatinine≤1.5 × ULN or creatinine clearance (either measured value or estimated value using the Cockcroft-Gault equation) >60ml/min.

Exclusion Criteria:

1. Has HER2-positive or indeterminate gastric cancer
2. Have multiple cancers
3. Have a current or past history of severe hypersensitivity to any other antibody products
4. Have concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease
5. Have a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging (preferably CT) or clinical findings
6. Have brain or meninx metastases. Patients may be randomized for the study if they are asymptomatic and require no treatment.
7. Have pericardial fluid, pleural effusion, or ascites requiring treatment
8. Have a history of uncontrollable or significant cardiovascular disease
9. Have systemic infection requiring treatment
10. Are contraindicated for paclitaxel
11. Has had prior treatment with:

    - Require or, within 28 days before treatment, have received systemic corticosteroids or immunosuppressants
12. Have undergone surgery (any surgery involving general anesthesia) within 28 days before study treatment
13. Have received radiotherapy for gastric cancer within 28 days before treatment or radiotherapy for bone metastases within 14 days before treatment
14. Have a positive test result for human immunodeficiency virus-1 (HIV-1) antibody,
15. Hepatitis B surface protein (HBs) antigen and HBV titer >2000 IU/ml (10,000 copy/ml), or hepatitis C virus (HCV) antibody positive result
16. Are pregnant or breastfeeding, or possibly pregnant
17. Has any unresolved ≥Grade 2 (per CTCAE v4.0) toxicity from previous anti-cancer therapy at the time of enrollment such as neuropathy, except alopecia or anemia
18. Have previously received nivolumab, anti-programmed cell death-1 (PD-1) antibody, anti-PD-L1 antibody, anti-programmed cell death-ligand 2 (PD-L2) antibody, anti-CD137 antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) antibody, or other therapeutic antibodies or pharmacotherapies for the regulation of T-cells
19. Are incapable of providing consent for specific reasons, such as concurrent dementia
20. Are otherwise inappropriate for this study in the investigator's or subinvestigator's opinion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
(Phase Ib) Maximum Tolerated dose (MTD) | 424 weeks
  Maximum Tolerated dose (MTD) as determined by Dose limiting Toxicity (DLT).
(Phase Ib) Recommended phase 2 dose | 424 weeks
  Recommended phase 2 dose as determined by Dose limiting Toxicity (DLT).
(Phase II) PFS | 424 weeks
  Progression-free survival (PFS): Defined as the time from start of study treatment until the date of objective disease progression or death (by any cause in the absence of disease progression) Progression is defined in accordance with the RECIST v1.1 criteria. PFS is defined as the interval between the date of first dose and the earliest date of disease progression or death due to any cause.

SECONDARY OUTCOMES:
OS | 24 weeks
  Overall Survival (OS): the time from the date of first dose and the date of death from any cause
ORR | 24 weeks
  Overall response rate (ORR): defined as the percentage of subjects with a confirmed CR or PR per RECIST v1.1 relative to the total number of subjects
DCR | 24 weeks
  Disease Control Rate (DCR): the proportion of randomized patients achieving a best overall response of CR, PR, or SD.
PFS | 24 weeks
  Progression-free survival (PFS): To evaluate the treatment effect of nivolumab and paclitaxel on progression-free survival (PFS) rate at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG RHA, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No